CLINICAL TRIAL: NCT03291574
Title: Effect of Perioperative Electroacupuncture After Gastrectomy for Gastric Cancer Patients on Rapid Rehabilitation: A Randomized Clinical Trial
Brief Title: Perioperative Electroacupuncture for Gastric Cancer Patients After Gastrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Chengfeng Wang, Director of Department of pancreatic and gastric Surgery, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LC2015L45
Record Dates: First submitted 2017-07-29; First posted 2017-09-25 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Acupuncture; Gastrointestinal Function
MeSH Terms: interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture group (Experimental): Acupuncture at Baihui, Nei guan, bilateral Zu sanli and bilateral Tian shu
  Interventions: Procedure: Electroacupuncture
- Sham electroacupuncture group (Placebo Comparator): Sham acupuncture at Baihui, Nei guan, bilateral Zu sanli and bilateral Tian shu
  Interventions: Procedure: Sham electroacupuncture

INTERVENTIONS:
Procedure: Electroacupuncture — Acupuncture at Baihui, Nei guan, bilateral Zu sanli and bilateral Tian shu.
  Arms: Electroacupuncture group
Procedure: Sham electroacupuncture — Sham acupuncture at Baihui, Nei guan, bilateral Zu sanli and bilateral Tian shu.
  Arms: Sham electroacupuncture group

SUMMARY:
Evaluate the effect of Perioperative Electroacupuncture on rapid rehabilitation for the gastric cancer patients after gastrectomy .

DETAILED DESCRIPTION:
The trial is funded by Cancer Foundation of China. The trial is prepared to be registered on the clinicaltrail.gov. Quality assurance plan: every participant is enrolled or excluded by two practiced investigators. And two investigators participated in all steps of the trail, including the record of the data, and the investigators will compare the data. If the data is consistent, the investigators would record the data; if not, the data would be checked and decided by the two investigators. All the steps and data are site monitored and audited by the workers of research and financial department of National Cancer Center/ Cancer Hospital, Chinese Academy of Medical Sciences. Data check: the investigators compare data entered into the registry against predefined rules for range or consistency with other data fields in the registry. Source data verification to assess the accuracy, completeness, or representativeness of registry data by comparing the data to external data sources, including medical records and electronic case report forms. Data dictionary that contains detailed descriptions of each variable used by the registry, including the source of the variable, coding information, and normal ranges if relevant.

Standard Operating Procedures to address registry operations and analysis activities, such as participants recruitment, data collection, data management, data analysis, reporting for adverse events, and change management. All registry operations would be done according to specific steps, and by two practiced investigators. Sample size assessment to specify the number of participants or participant years necessary to demonstrate an effect. According to the formula to differ advantages and disadvantages, the investigators need at least 70 participants to take part in the trail.

The investigators can recruit about 35 participants every year according to previous experiences, so the investigators should recruit at least for two years. Plan for missing data: the investigators would collect as much data as possible, and the investigators exclude the participants who cannot cooperate on recruitment. And the investigators manage situations according to statistical principles where variables are reported as missing, unavailable, "non-reported," uninterpretable, or considered missing because of data inconsistency or out-of-range results. Statistical analysis plan: Kaplan-Meier method would be used to analyze the difference of survival time between the two groups, and the local control rate of the two groups would be compared by chi square test. Statistical analyses would be performed by using IBM SPSS Statistics(version 20; IBM, Chicago, USA). The level of significance is defined as P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with gastric cancer who undergoing gastrectomy.
2. The life expectancy will be more than 3 months.
3. Voluntary participation, Signing informed consent and have good compliance.

Exclusion Criteria:

1. Patient who has a history of abdominal surgery, radiotherapy, and chemotherapy.
2. Patient who combined with abdominal lymph node metastasis or distant organ metastasis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2017-07-29 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal function score | day 1 after surgery
  Using scale to evaluate the function of gastrointest after surgery
Gastrointestinal function score | day 3 after surgery
  Using scale to evaluate the function of gastrointest after surgery
Gastrointestinal function score | day 5 after surgery
  Using scale to evaluate the function of gastrointest after surgery
Gastrointestinal function score | day 7 after surgery
  Using scale to evaluate the function of gastrointest after surgery

SECONDARY OUTCOMES:
Physical fitness index | day 1 after surgery
  The recovery of physical fitness index
Physical fitness index | day 3 after surgery
  The recovery of physical fitness index
Physical fitness index | day 5 after surgery
  The recovery of physical fitness index
Physical fitness index | day 7 after surgery
  The recovery of physical fitness index

CONTACTS AND LOCATIONS:
Overall Officials: chenefeng Wang, B.A, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Qiu G, Huang T, Lu Y, Zhang L, Zhao Y, Yuan Y, Ren H, An J, Zhou J, Li R, Du Y, Wang T, Wang P, He F, Ding Y, Zhang J, Han B, Lan Z, Qi S, Li Z, Gao J, Gu Z, Sun Y, Bai X, Aimaiti S, Chu Y, Wang C. Perioperative Electroacupuncture Can Accelerate the Recovery of Gastrointestinal Function in Cancer Patients Undergoing Pancreatectomy or Gastrectomy: A Randomized Controlled Trial. Evid Based Complement Alternat Med. 2021 Mar 31;2021:5594263. doi: 10.1155/2021/5594263. eCollection 2021. PMID 33859707